CLINICAL TRIAL: NCT06985875
Title: Clinical Trial for the Evaluation of the Safety and Efficacy of a Moisturizing Solution With Hyaluronic Acid Drop 0.4%
Brief Title: Clinical Trial for the Evaluation of Safety and Efficacy of Drop 0.4%
Acronym: DROP04
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avizor SA (Industry)
Collaborators: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IOBA-Avizor 001-2024
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Eye Dryness
Keywords: contact lens, dry eye
MeSH Terms: conditions — Xerophthalmia; Dry Eye Syndromes | interventions — Preservation, Biological

STUDY DESIGN:
Intervention Model Description: Both Arms receive both Investigational product and comparator in a crossover design. Randomization determines the order of administration. A washout period between both treatments is performed.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Product and comparator have the same external and physical characteristics and the label is the same for both products except for expiry date
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contact lens users with eye dryness (Other): Contact lens users that have eye dryness symptoms. Both treatments will be administered, as it is a crossover study.
  Interventions: Device: Multidose mosturizing solution DROP 0.4%; Device: Multidose mosturizing solution Avizor Eye Drops 0.2% Preserved
- Non contact lens user with eye dryness (Other): Non contact lens patients with eye dryness symptoms. Both treatments will be administered, as it is a crossover study.
  Interventions: Device: Multidose mosturizing solution DROP 0.4%; Device: Multidose mosturizing solution Avizor Eye Drops 0.2% Preserved

INTERVENTIONS:
Device: Multidose mosturizing solution DROP 0.4% — Ophthalmic mosturizing solution to be administered 1-4 times per day in both eyes
Device: Multidose mosturizing solution Avizor Eye Drops 0.2% Preserved — Ophthalmic mosturizing solution to be administered 1-4 times per day in both eyes

SUMMARY:
The aim of the trial is to compare the safety and efficacy of the moisturizing solution DROP 0.4% with the moisturizing solution AVIZOR EYE DROPS 0.2% PRESERVED in relieving the symptoms of dry eye over one month of use.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female, aged 18 years or older, capable of freely providing informed consent for participation in the study.
* Signed informed consent form prior to any study-related tests.
* Signed data protection form prior to any study-related tests.

Additionally, for Group 1 (Non contact lens users)

* Ocular surface disease index (OSDI) ≥ 13
* No use of contact lenses in the past month and not planning to use them during the study period.

Additionally, for Group 2 (contact lens users)

* Contact lens dry eye questionnaire (CLDEQ-8) ≥ 12
* Contact lens (CL) use with a habitual minimum use of 4 days per week and 4 hours per day in the past month.

EXCLUSION CRITERIA:

* Any active ocular surface disease except for dry eye disease.
* Severe dry eye, defined as meeting at least one of the following criteria in at least one eye:

  * Corneal fluorescein staining ≥ 4 on the Oxford scale (0-5).
  * Conjunctival lissamine green staining ≥ 4 on the Oxford scale (0-5).
  * Schirmer test value ≤ 2 mm.
  * Tear stability (BUT) of 0 seconds.
* History of ocular surgery in the last 3 months or refractive corneal surgery in the last 6 months.
* History of herpetic keratitis or uveitis.
* History of severe ocular infections or inflammation in the 6 months prior to the study.
* History of allergies affecting the ocular surface during the study period.
* Patients who have started or are expected to modify the use of the following topical medications during the study (except for artificial tears/moisturizing and lubricating solutions):

  * Calcineurin inhibitors (cyclosporine, tacrolimus, etc.) in the 12 weeks prior to the study.
  * Corticosteroids or non steroid anti-inflammatory drugs (NSAID) in the 4 weeks prior to the study.
  * Blood-derived treatments (autologous serum, enriched plasma, etc.), insulin, or amniotic preparations in the week prior to the study.
* Use of systemic medication with potential effects on the tear film that has been started or modified in the last month or is expected to change during the study.
* Known sensitivity or intolerance to any of the products used in the study.
* Subjects with clinically relevant or uncontrolled systemic diseases in the last 3 months that may interfere with study assessments or outcomes.
* Pregnancy or breastfeeding. Lack of effective contraceptive methods in women of childbearing potential.
* Participation in a clinical trial within the last 30 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in eye dryness symptoms | 1 month
  Changes in ocular symptoms (measured with Contact lens dry eye questionnaire and/or change in the frequency and intensity of dry eye symptoms (measured with a Visual analogue scale from 0 to 10). For contact lens users
Changes in eye dryness symptoms | 1 month
  Changes in ocular symptoms (measured with Ocular surface disease index and/or change in the frequency and intensity of dry eye symptoms (measured with a Visual analogue scale from 0 to 10). For non contact lens users
Changes in best corrected visual acuity (safety outcome) | 1 month
  Best corrected visual acuity tested with ETDRS (early treatment for diabetes retinopathy study).
Ocular and peri orbital adverse events | 1 month
  All local adverse events reported
Serious adverse events | 1 month
  All local and systemic serious adverse events

SECONDARY OUTCOMES:
Stability of the tear film | 1 month
  Measurement of tear film stability by Non-Invasive Break-Up Time (NIBUT).
Ocular surface response to treatment - Oxford Scale (0 (Better) to 5 (Worse)) | 1 month
  Corneal staining with fluorescein, green lissamine and conjunctival hyperemia
Tear evaporation | 1 month
  Assessed by evaporimetry
Number of instillations per product | 1 month
  Comparison between the number of intimations of both products
User satisfaction with the product | 1 month
  Numerical scale from 1 to 10

IPD SHARING:
Plan to Share IPD: No